CLINICAL TRIAL: NCT01191502
Title: Comparative Study of Photopic and Mesopic Distance Intermediate and Near Visual Acuity, and Spectacle Independence With Binocular Implantation of the Tecnis Multifocal (TMF) Intraocular Lens or Crystalens HD (CHD) Intraocular Lens
Brief Title: Comparative Study of Photopic and Mesopic Distance, Intermediate and Near Visual Acuity, and Spectacle Independence
Status: Completed | Type: Observational
Sponsor: Innovative Medical (Industry)
Responsible Party: Mark Packer, Oregon Health & Sciences University
Other Study IDs: TMF-09-002
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Visual Acuity
Keywords: Patients who have had binocular implantation of the Tecnis Multifocal IOL or the Crystalens™ HD Accommodating IOL.

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TECNIS MULTIFOCAL (TMF) INTRAOCULAR LENS
- CRYSTALENS HD (CHD) INTRAOCULAR LENS

SUMMARY:
The purpose of this study is to evaluate visual acuity in different lighting conditions (daylight and night time) and distances (distance, near and intermediate), and the independence of glasses, in patients who have had binocular implantation of the Tecnis Multifocal IOL or the Crystalens™ HD Accommodating IOL.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Status post bilateral cataract or refractive lens surgery (with or without LRI) and implantation of Tecnis™ Multifocal IOL or Crystalens™ HD Accommodating IOL
* Best-corrected ETDRS equivalent visual acuity of 20/30 or better in each eye
* Naturally dilated pupil size (in dim light) > 3.5 mm (with no dilation medications) for both eyes
* Clear intraocular media (no posterior capsular opacification, or status post YAG capsulotomy)
* Availability, willingness, and sufficient cognitive awareness to comply with examination procedures

Exclusion Criteria:

* Ocular disease which could potentially limit uncorrected visual acuity or visual performance.
* Use of systemic or ocular medications that may affect visual outcomes
* Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus, immunocompromised, etc.)
* Uncontrolled systemic or ocular disease
* History of ocular trauma
* History of ocular surgery other than that required for inclusion in this study
* Amblyopia or strabismus
* Known pathology that may affect visual acuity; particularly retinal changes that affect vision (macular degeneration, cystoid macular edema, proliferative diabetic retinopathy, etc.)
* Diagnosed degenerative visual disorders (e.g. macular degeneration, or other retinal disorders) that are predicted to cause future acuity losses to a level of worse than 20/30
* Subjects who may be expected to require retinal laser treatment or other surgical intervention
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome)
* Pupil abnormalities (non-reactive, tonic pupils or abnormally shaped pupils)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Evaluate visual acuity in different lighting conditions (daylight and night time) and distances (distance, near and intermediate), and the independence of glasses, in patients who have had binocular implantation of the Tecnis Multifocal IOL or the Crystalens™ HD Accommodating IOL.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Manifest refraction (monocular) | 1 year
Uncorrected visual acuity (UCVA) ETDRS testing at distance, intermediate and near in photopic lighting (monocular and binocular) | 1 year
Best distance-corrected visual acuity (BDCVA) ETDRS testing at distance, intermediate and near in photopic lighting (monocular and binocular) | 1 year
Uncorrected visual acuity (UCVA) ETDRS testing at distance, intermediate and near in mesopic lighting (monocular and binocular) | 1 year
Best distance-corrected visual acuity (BDCVA) ETDRS testing at distance, intermediate and near in mesopic lighting (monocular and binocular) | 1 year
Photopic and mesopic pupillometry | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Sciences University, Eugene, Oregon, United States